CLINICAL TRIAL: NCT01032980
Title: Post Authorization Safety Study of the Intramuscular Inactivated, Split Virion Pandemic A/H1N1 Influenza Vaccines in Children Aged Over 2 Months and in Adult Populations
Brief Title: Post Authorization Safety Study of the Pandemic A/H1N1 Influenza Vaccines in Children and Adults
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: GPF11; UTN: U1111-1112-2748 (Other: WHO)
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Influenza; Swine-Origin A/H1N1 Influenza Virus
Keywords: HUMENZA; PANENZA; Influenza; Swine-Origin Influenza A H1N1 Virus; Influenza virus vaccines
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HUMENZA Vaccine Group: Participants vaccinated with HUMENZA according to the recommendations provided in the product leaflet and local recommendations.
- PANENZA Vaccine Group: Participants vaccinated with PANENZA according to the recommendations provided in the product leaflet and local recommendations.

SUMMARY:
This study is designed to assess the safety of the approved and licensed HUMENZA (adjuvanted A/H1N1 pandemic influenza vaccine) and PANENZA (non-adjuvanted A/H1N1 pandemic influenza vaccine) to meet regulatory requirements for post-marketing safety monitoring.

Primary objective:

To describe the incidence of serious adverse events and adverse events of special interest (AESIs) after HUMENZA or PANENZA administration throughout the study in different age groups.

Secondary objective:

To describe the incidence of non-serious cutaneous allergic reactions after HUMENZA or PANENZA administration in different age groups up to 21 days after the last vaccination.This study is designed to assess the safety of the approved and licensed HUMENZA (adjuvanted A/H1N1 pandemic influenza vaccine) and PANENZA (non-adjuvanted A/H1N1 pandemic influenza vaccine) to meet regulatory requirements for post-marketing safety monitoring.

DETAILED DESCRIPTION:
All participants will be vaccinated with study vaccines (1 or 2 doses) at the start of the study and will be monitored for safety for up to 6 months after the last vaccination.

ELIGIBILITY:
Inclusion Criteria :

* Aged 2 months and above on the day of inclusion
* Having received HUMENZA or PANENZA
* Provision of the Contact Order Form (COF) signed by the participant or the participant's parent(s)/guardians(s)
* Participant or the participant's parent(s)/legal representative(s) are able to attend all scheduled visits and to comply with all study procedures

Exclusion Criteria :

* Participant previously vaccinated with another A/H1N1 pandemic vaccine

Min Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be vaccinated with HUMENZA or PANENZA according to the recommendations provided in the product leaflet and local recommendations.
  The HUMENZA Group will be divided in 6 defined age groups; the PANENZA Group will be divided into 2 defined age groups.
Sampling Method: Non-Probability Sample
Enrollment: 3934 (Actual)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Safety: To provide information concerning the safety of HUMENZA and PANENZA vaccines. | 21 days post-vaccination and entire study duration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (5):
- France (5):
  - Bordeaux
  - Lille
  - Lyon
  - Marseille
  - Paris

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com